CLINICAL TRIAL: NCT07131917
Title: Feasibility, Safety and Clinical Impact of Bedside Microenvironmental Monitoring in Infected Walled-Off Pancreatic Necrosis During Standard Percutaneous Drainage
Brief Title: Bedside Monitoring of Microenvironmental Changes in Infected Pancreatic Collections
Acronym: WOPN-MONITOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Harazim (Other)
Responsible Party: Sponsor-Investigator, Martin Harazim, Principal Investigator, Department of Gastroenterology and Intensive Care Medicine, Brno University Hospital
Organization: Brno University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WOPN-MONITOR-001
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pancreatitis; Walled Off Pancreatic Necrosis
Keywords: pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: All enrolled participants undergo standard percutaneous drainage of infected WOPN. A single-arm study assesses feasibility and clinical impact of adding bedside microenvironmental monitoring using a miniaturized sensor probe temporarily inserted into the collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bedside Microenvironment Monitoring Arm (Experimental): Participants in this arm will undergo standard percutaneous drainage of infected walled-off pancreatic necrosis (WOPN) as per clinical indication. In addition, a sterile, biocompatible micro-monitoring probe will be temporarily introduced into the collection to measure local microenvironmental parameters. Measurements will be performed intermittently or continuously for up to 72 hours without compromising drainage function. No investigational drug or therapeutic intervention is administered.
  Interventions: Device: Miniaturized Intracavitary Monitoring Probe

INTERVENTIONS:
Device: Miniaturized Intracavitary Monitoring Probe — A sterile, miniaturized, biocompatible monitoring probe (≤1.5 mm diameter) is temporarily introduced into the cavity of an infected walled-off pancreatic necrosis (WOPN) during standard percutaneous drainage. The device is designed to measure local microenvironmental parameters in situ, such as acidity and related indicators, without interfering with fluid evacuation. Measurements are performed intermittently or continuously for up to 72 hours and are used solely for observational purposes. This intervention is distinct from standard WOPN management, as it allows real-time assessment of local physicochemical conditions, which are not accessible through systemic biomarkers or imaging alone.

SUMMARY:
This pilot clinical study aims to assess the feasibility and clinical relevance of bedside monitoring of microenvironmental conditions within infected walled-off pancreatic necrosis (WOPN).

WOPN is a serious complication of acute pancreatitis, often associated with infection, organ failure, and the need for drainage or surgical intervention. Although infection is a key factor in prognosis, little is known about the local chemical environment inside the infected collections.

In this study, a sterile, miniaturized probe will be temporarily introduced into the necrotic cavity during standard percutaneous drainage. The goal is to record local microenvironmental parameters (such as acidity or related values) and monitor their changes over time.

By comparing these values with clinical data (e.g., inflammatory markers, microbiology, need for surgery), the study aims to determine whether such measurements can provide additional information about infection severity and treatment response.

The study does not involve any experimental treatment. All patients will receive standard medical care, including antibiotics, imaging, and drainage according to international guidelines.

Participation is voluntary. Only patients who provide informed consent will be enrolled.

DETAILED DESCRIPTION:
Background:

Infected walled-off pancreatic necrosis (WOPN) represents a critical complication of acute necrotizing pancreatitis. Management typically includes antibiotics and step-up interventional drainage. However, decision-making is often based on indirect systemic markers, and very little is known about the actual in situ microenvironmental conditions (e.g., pH, oxygenation, redox status) inside the necrotic cavity.

Rationale and Innovation:

The metabolic and microbiological activity within infected WOPN likely alters the local chemical environment, particularly in terms of acidity and anaerobic conditions. These changes may influence pathogen virulence, host immune response, and - importantly - the stability and efficacy of administered antibiotics. There is currently no standard method for directly monitoring these local parameters at the bedside. This pilot study explores the feasibility and potential clinical value of such monitoring.

Objective:

To determine whether bedside microenvironmental monitoring inside infected WOPN is feasible, safe, and potentially useful for clinical decision-making.

Methods:

This is a single-arm, prospective, interventional feasibility study. Patients with clinically confirmed infected WOPN undergoing standard percutaneous drainage will be offered participation. A sterile, biocompatible mini-probe (≤1.5 mm diameter) will be introduced into the collection during drainage and used to monitor selected parameters (e.g., pH) intermittently or continuously for up to 24-72 hours. The sensor will be removed safely without compromising drainage.

Data will be collected on insertion feasibility, measurement quality, patient tolerance, and any complications. Clinical parameters (CRP, PCT, SOFA score), microbiology, and clinical outcomes (resolution of infection, need for surgery, mortality) will be tracked and compared with measured values.

Outcomes:

Primary outcomes include the feasibility of safe insertion and measurement, and preliminary correlation with infection severity and clinical course. Secondary outcomes include association of monitored values with microbiology, organ dysfunction, and treatment response.

Future Direction:

If successful, this study will lay the groundwork for larger observational trials and possibly interventional studies using pH- or microenvironment-guided therapy (e.g., antibiotic selection or early intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of walled-off pancreatic necrosis (WOPN) confirmed by imaging (CT, MRI, or EUS)
* Clinical suspicion or confirmation of infection in WOPN (e.g., fever, elevated inflammatory markers, positive culture)
* Planned percutaneous drainage as part of standard care
* Ability to provide informed consent (or surrogate consent where applicable)

Exclusion Criteria:

* Coagulopathy not correctable prior to intervention (e.g., INR > 2.0 or platelets < 50×10⁹/L)
* Known allergy or hypersensitivity to materials used in the monitoring probe
* technical limitations precluding safe probe insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Safety of Intracavitary Monitoring During Percutaneous Drainage of Infected WOPN | From Day 0 (drainage procedure) to Day 3 or removal of the probe, whichever occurs first
  Successful placement, function, and removal of the miniaturized monitoring probe during standard percutaneous drainage of infected WOPN. Feasibility is defined as the ability to insert the probe without interrupting drainage, record interpretable data for at least 24 hours, and remove the device without adverse events. Safety is assessed by the absence of procedure-related complications, such as bleeding, infection exacerbation, or drainage dysfunction related to the monitoring device.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
This is a single-center pilot study with a limited sample size and exploratory objectives. The decision to share individual participant data (IPD) will depend on the quality, completeness, and generalizability of the collected data, as well as institutional and ethical considerations regarding data anonymization and reuse. A data sharing plan may be developed in future phases of research if the findings support broader dissemination.

REFERENCES:
- See also: Related Info — https://www.fnbrno.cz